CLINICAL TRIAL: NCT06288672
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of Patch Test-Guided Type 4 Food Allergen Dietary Avoidance for Irritable Bowel Syndrome
Brief Title: IBS Skin Patch Test Food Allergy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBS-80, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1003A
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; IBS; FODMAP; low FODMAP; IBS diet; IBS food allergy; IBS solution; IBS treatment; IBS foods; low FODMAP diet; IBS evaluation; irritable bowel syndrome treatment; irritable bowel syndrome management; IBS cause; irritable bowel syndrome pathogenesis; irritable bowel syndrome evaluation; IBS pathogenesis
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants with IBS are patch tested to 80 type 4 food allergens. Those with questionable or positive patch test reactions are randomized to follow a patch test-directed avoidance diet or a sham diet (avoidance of foods to which the patch tests showed no reaction) for 16 weeks. Upon conclusion of the avoidance diet, participants complete a brief questionnaire to assess their response to the avoidance diet.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The true or sham avoidance diet for each participant is randomly assigned by the study administrator. Assignments will not be made available to participants until after their study completion or to investigators until all 250 participants have completed the study and the results have been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True avoidance diet (Active Comparator): Food patch test-directed avoidance diet for 16 weeks where participant avoids avoid eating the food(s) to which they are allergic
  Interventions: Other: True avoidance diet
- Sham avoidance diet (Sham Comparator): Avoidance diet for 16 weeks of randomly selected foods to which the patch testing did not show an allergy
  Interventions: Other: Sham avoidance diet

INTERVENTIONS:
Other: True avoidance diet — Food patch test-directed avoidance diet for 16 weeks where participant avoids avoid eating the food(s) to which they are allergic
  Arms: True avoidance diet
Other: Sham avoidance diet — Avoidance diet for 16 weeks of randomly selected foods to which the patch testing did not show an allergy
  Arms: Sham avoidance diet

SUMMARY:
Participants with IBS are skin patch tested (no needles) to 80 different foods and food additives, compounded for patch testing, in search of food allergies. The testing requires 3 office visits within a 4 or 5 day period. The patches are taped to the back at Visit #. At Visit #2 48 hours later, the patches are removed from the skin and the outside border of each patch is marked with a felt tip marker. At Visit #3 (final visit) 1 or 2 days later, the patch test reading is performed by the doctor-investigator. An allergy is identified as a small red mark where the food was in contact with the skin for 48 hours. Those participants found to have food allergies are then placed on an avoidance diet (no calorie restriction) for 16 weeks where they either avoid eating the food(s) to which they are allergic (the "true" avoidance diet) or food(s) to which the testing did not show an allergy (this is called the "sham" avoidance diet). There is a 50/50 chance of going on either avoidance diet. The avoidance diet is assigned in such a way that neither the participant or the doctor-investigator knows which diet is being followed. After the 16 weeks, the participants answers a brief online questionnaire that asks about the IBS symptoms while following the avoidance diet. After the 16 week avoidance diet and final questionnaire are completed, those participants who were on the sham diet will be told of their true food allergies which they may try avoiding on their own.

DETAILED DESCRIPTION:
See above. When all 250 study participants have finished all parts of the study, the results will be made known to the doctor-investigators for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Irritable bowel syndrome diagnosed by a primary care provider, gastroenterologist or allergist; or
2. meeting the Rome IV IBS diagnostic criteria by history and having suboptimally or poorly controlled IBS symptoms.

Exclusion Criteria:

1. Under age 18 years
2. Pregnant
3. Severe rash
4. Receiving any cortisone-containing or any of the following immunosuppressive medications within two weeks prior to patch testing or plan to do so any time during the study: cyclosporine, mycophenylate mofetil, azathioprine, tacrolimus or others within these classes of medications)
5. Incapable of completing all parts of the 18-week screening period and study, including following the dietary instructions and completing all text or email questionnaires
6. Exposure of back to the sun in the 2 weeks prior to patch testing Unable or unwilling to discontinue the low FODMAP diet, if relevant, starting 1 week prior to the study and for the study duration

8) Refusal to shave back hair, if relevant 9) Receiving pharmacologic therapy for IBS that has been started or changed within 30 days of study enrollment 10) Non-English speaking 11) Unable to provide written informed consent 12) Have a history of gastrointestinal disease including celiac disease, cirrhosis, gastrointestinal malignancy, inflammatory bowel disease, or diverticulitis, active within the prior 2 years. 13) Have a history of gastrointestinal surgery (except appendectomy and cholecystectomy or gallbladder removal >6 months ago) 14) Have poorly controlled psychiatric disease such as severe depression (with or without suicidal ideation), severe anxiety, schizophrenia, dementia 15) Have excessive alcohol intake (more than 1 drink per day for females and 2 drinks per day for males) 16) Use illicit substances 17) Use high-dose opiates 18) Severe allergy to adhesive tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-Avoidance Diet Relative IBS Symptom Global Assessment | Questionnaire to be completed promptly after completion of 16 week avoidance diet.
  Participant global assessment of IBS symptoms compared to the three months prior to entering study, assessed by a post-avoidance diet questionnaire. The assessment is a 7 point Likert scale with 1=substantially improved; 2=moderately improved; 3=slightly improved; 4=no change; 5=slightly worse; 6=moderately worse; 7=substantially worse

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Stierstorfer, MD, Principal Investigator — North Wales Dermatology, PLLC
Locations (2):
- United States (2):
  - North Wales Dermatology, PLLC, North Wales, Pennsylvania
  - Shepherd Allergy, Barboursville, West Virginia

REFERENCES:
- [Background] Shin GH, Smith MS, Toro B, et al. Utility of food patch testing in the evaluation and management of irritable bowel syndrome. Skin. 2018;2:1-15.
- [Result] Stierstorfer MB, Toro B. Patch Test-Directed Dietary Avoidance in the Management of Irritable Bowel Syndrome. Cutis. 2021 Aug;108(2):91-95. doi: 10.12788/cutis.0321. PMID 34735319
- [Result] Stierstorfer MB, Sha CT, Sasson M. Food patch testing for irritable bowel syndrome. J Am Acad Dermatol. 2013 Mar;68(3):377-84. doi: 10.1016/j.jaad.2012.09.010. Epub 2012 Oct 24. PMID 23102771